CLINICAL TRIAL: NCT05847049
Title: Influence of Combined Eplerenone , Intravitreal Aflibercept and Topical Nepafenac Therapy on Serous Foveal Detachment in Central Serous Chorioretinopathy (CSCR)
Brief Title: Eplerenone, Aflibercept and Topical Nepafenac Serous Foveal Deta Chment in Central Serous Chorioretinopathy
Acronym: CSCR
Status: Completed | Type: Observational
Sponsor: Dar El Oyoun Hospital (Other)
Responsible Party: Principal Investigator, Wael Ahmed Ewais, Associate professor of ophthalmology, Dar El Oyoun Hospital
Other Study IDs: N-20-2023
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Eplerenone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Eplerenone , Intravitreal Aflibercept and Topical nepafenac therapy — Eplerenone , Intravitreal Aflibercept and Topical nepafenac therapy

SUMMARY:
describing the influence of; combined Eplerenone, intravitreal Aflibercept, and topical Nepafenac; on serous foveal detachment in eyes with CSCR

DETAILED DESCRIPTION:
Retrospective Review of records of eyes with Central serous chorioretinopathy (CSCR) that have been treated in the period between 2015 and 2021

After checking inclusion and exclusion criteria; we will enroll all cases that have been treated by the combination of eplerenone, intravitreal aflibercept and topical nepafenac.

Investigators collected and recorded the following data:

* Age
* Gender
* Systemic hypertension (present or not)
* Smoking (Yes / No)
* Best corrected visual acuity (BCVA) (baseline, final)
* Central macular thickness (CMT) (baseline, final)
* Serous detachment Height (SDH) (baseline, final)
* Duration of Follow-up ( in months)

ELIGIBILITY:
Inclusion Criteria:

* CSCR eyes treated by combination of Eplerenone, Aflibercept and Nepafenac.

Exclusion Criteria:

* • CSCR treated by other modalities

  * CSCR treated by just 1 or 2 components of :Eplerenone, Aflibercept and Nepafenac

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eyes with Central serous chorioretinopathy (CSCR) that have been treated in the period between 2015 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Change in central macular thickness (CMT ) in microns | (baseline, 6 months)
  reduction in CMT after therapy
Change in serous detachment height (SDH) in microns | (baseline, 6 months)
  reduction in SDH after therapy

SECONDARY OUTCOMES:
Change in BCVA | (baseline, 6 months)
  number of lines of improvement in BCVA after therapy
Duration of Follow-up ( in months) | (baseline, 6 months)
  Duration of Follow-up ( in months)
Complications (Eplerenone, Aflibercept, and nepafenac) | (baseline, 6 months)
  present or absent

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No